CLINICAL TRIAL: NCT04387162
Title: One Treatment, Multiple Targets: Prism Adaptation and Left Brain Stroke Rehabilitation
Brief Title: Prism Adaptation in Left Brain Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B3474-P; RX003474-01 (Other Grant/Funding Number: VAORD)
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Aphasia; Spatial Neglect; Stroke
Keywords: aphasia; spatial neglect; rehabilitation
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: Multiple baseline, delayed treatment design
Who Masked: Outcomes Assessor
Masking Description: Neurologist will conduct blinded classification of "frontal" or "nonfrontal" lesions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate (Experimental): Participants will enter treatment after one week baseline
  Interventions: Behavioral: Prism Adaptation Treatment
- Delayed (Experimental): Participants will enter treatment after two week baseline
  Interventions: Behavioral: Prism Adaptation Treatment

INTERVENTIONS:
Behavioral: Prism Adaptation Treatment — Spatial retraining treatment

SUMMARY:
Of the 15,000 Veterans who are hospitalized for stroke each year more than half experience spatial and motor impairments and pain. Spatial-motor-sensory problems limit functioning and independence, which is costly to Veterans, their families, and society. Currently, spatial-motor-sensory problems are targeted using different treatments. However, there is a treatment that has shown promise in simultaneously targeting spatial function, motor function and pain in right-brain stroke. The investigators propose to investigate the feasibility of using adapted spatial-motor sensory assessment and treatment procedures for Veterans with left-brain stroke who have language and cognitive impairment. The next step will be to conduct a large-scale study focused on this multi-target treatment for more efficient and effective stroke rehabilitation. The investigators expect this line of research to increase functioning, independence and quality of life in Veteran stroke survivors.

DETAILED DESCRIPTION:
The functional disability experienced by Veterans after stroke, and the limited rehabilitation resources available, highlight the importance of identifying feasible treatments acting on more than one recovery target. Currently, there are separate and modality-specific treatment pathways for cognitive and motor impairments. These modality-specific treatment pathways lead to fragmentation of care, and under-identification and under-treatment of invisible disabilities, such as spatial neglect, aphasia and pain. The result is longer hospital stays, greater risk of falls, and poor functional outcomes. Employing a treatment that simultaneously addresses multiple targets will ensure that the investigators provide the needed care for >50% of post-stroke Veterans who have both visible and invisible disabilities, during the critical post-acute period of recovery.

Prism adaptation treatment (PAT) is a 10-day regimen reported to be inexpensive, replicable and effective for treatment of spatial neglect, and studies have demonstrated that it also enhances everyday activities and motor recovery and reduces chronic post-stroke pain in patients with right brain stroke. Additionally, brain mapping methods have shown that in patients with right brain stroke, those with frontal lesions respond optimally to PAT. No studies have investigated PAT in left-brain stroke patients with language and cognitive impairment. To address this research gap, the investigators will address the following aims:

Aim 1: To demonstrate the feasibility of adapted PAT procedures in patients with aphasia and memory impairment. .

Aim 2: To demonstrate the feasibility of adapted methods for assessing spatial and motor function and pain in patients with aphasia and memory impairment.

Aim 3: To demonstrate the feasibility of using information about lesion location from the radiology report to classify frontal vs. nonfrontal lesions.

ELIGIBILITY:
Inclusion Criteria:

* 1-3 months post-stroke, entering outpatient treatment
* proficient English speakers
* experiencing moderate functional disability as measured by Functional Independence Measure (FIM), observational or telephone-administered FONE-FIM
* experiencing aphasia as determined by a Western Aphasia Battery Aphasia Quotient and memory impairment as determined by the Brief Visuospatial Memory Test- Revised, the Hopkins Verbal Learning Test- Revised or digit span forward and backward
* able to provide informed consent to participate, using aphasia-accessible process, as needed.

Exclusion Criteria:

* History of brain conditions other than left brain stroke, including clinical right brain pathology.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Rodriguez, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight participants were consented into the study to complete screening procedures and ultimately did not meet eligibility criteria. These eight participants were not assigned to a study group.
Period: Overall Study
Arm/Group | Immediate | Delayed
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate | Delayed | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (9.1) | 53.5 (3.5) | 62.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire
Description: Assessment of satisfaction and perceived value of Prism Adaptation Treatment; scores range from 8-32, with higher scores indicating greater satisfaction
Time Frame: Immediately following the two-week treatment (study week 3 in immediate group, study week 5 in delayed group)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
score on a scale | 32 (0) | 27 (4.2)

2. Primary Outcome: Credibility/Expectancy Questionnaire
Description: Assessment of whether Prism Adaptation Treatment is believable, convincing and logical (credibility) and the expectations for treatment-induced improvement (expectancy); two rating scales with one scale ranging from 1-9 and from 0%-100%, with higher scores indicating greater credibility and expectancy.
Time Frame: Immediately following the two-week treatment (study week 3 in immediate group, study week 5 in delayed group)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
score on a scale
  Credibility | 6.2 (1.6) | 8.0 (.89)
  Expectancy | 56.7 (30.6) | 75.0 (7.1)

3. Primary Outcome: Barthel Index
Description: Assessment of functional disability by activities of daily living; scores range from 0-100, with higher score indicating greater independence and less functional disability
Time Frame: Weekly from baseline to follow-up (study week 7); baseline to immediate post-treatment (study week 3 in immediate group, study week 5 in delayed group), baseline to two weeks post-treatment (study week 7)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 70.8 (23.5) | 86.9 (10.9)
  Immediate Post-Treatment | 75.0 (22.9) | 82.5 (10.6)
  Two Weeks Post-Treatment | 71.7 (24.7) | 85.0 (7.1)

4. Primary Outcome: Functional Independence Measure
Description: Assessment of cognitive and motor function; scores range from 18-126, with a higher score indicating greater functional independence
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 88.2 (18.9) | 97.7 (9.1)
  Immediate Post-Treatment | 94.7 (21.7) | 98.5 (13.4)
  Two Weeks Post-Treatment | 95.0 (20.9) | 99.5 (13.4)

5. Primary Outcome: Behavioral Inattention Test- Conventional Subtest
Description: Assessment of spatial neglect; scores range from 0-146, with lower scores indicating more severe spatial neglect
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 115.3 (45.7) | 120.4 (5.3)
  Immediate Post-Treatment | 127.6 (24.9) | 119.0 (19.8)
  Two Weeks Post-Treatment | 127.3 (26.3) | 123.5 (3.5)

6. Primary Outcome: Catherine Bergego Scale Via the Kessler Foundation Neglect Assessment Process
Description: Assessment of spatial neglect; scores range from 0-30, with higher scores indicating more severe spatial neglect
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 3.6 (2.6) | 3.2 (2.4)
  Immediate Post-Treatment | 1.5 (2.6) | 1.5 (2.1)
  Two Weeks Post-Treatment | 1.5 (2.6) | 2.5 (3.5)

7. Primary Outcome: Wolf Motor Function Test
Description: Assessment of motor function; scores range from 0-75, with higher scores indicating less impairment in motor function
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 35.5 (30.7) | 54.3 (22.8)
  Immediate Post-Treatment | 35.7 (34.2) | 63.0 (14.1)
  Two Weeks Post-Treatment | 35.0 (34.7) | 65.0 (12.7)

8. Primary Outcome: Defense and Veterans Pain Rating Scale
Description: Assessment of pain; scores range from 0-10, with higher scores indicating more severe pain
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 0.5 (0.84) | 3.7 (2.2)
  Immediate Post-Treatment | 0.0 (0.0) | 3.5 (2.8)
  Two Weeks Post-Treatment | 0.7 (1.2) | 1.5 (2.1)

9. Primary Outcome: Classification of Lesion Location
Description: Assessment of whether lesion is "frontal" or "nonfrontal"
Time Frame: Baseline
Population: Unable to obtain records to complete this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of study entry until the end of study participation, an average of 2 months
Arm/Group | Immediate | Delayed
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
Significant issues were encountered with study recruitment. Screen fail rate was higher than anticipated. This resulted in a very small sample size. Data should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT04387162/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT04387162/ICF_001.pdf